CLINICAL TRIAL: NCT01917318
Title: A Double-Blind, Placebo-Controlled Random Order Crossover Study of Iloperidone for Symptoms of Arousal in PTSD Including Insomnia and Irritability.
Brief Title: Iloperidone for Symptoms of Arousal in Post Traumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment challenges - Single participant discontinued after placebo, no relevant outcome measure data was recorded.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-0207; IIRP-1371 (Other: Novartis pharmaceuticals)
Record Dates: First submitted 2013-07-31; First posted 2013-08-06 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post traumatic stress disorder; Treatment of post traumatic stress disorder; Symptoms of arousal in post traumatic stress disorder; Iloperidone in post traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — iloperidone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iloperidone / Placebo (Experimental): During 1st treatment period subjects will receive iloperidone. During 2nd treatment period subjects will receive placebo.
  Interventions: Drug: Iloperidone; Drug: Placebo
- Placebo / Iloperidone (Experimental): During 1st treatment period subjects will receive placebo. During 2nd treatment period subjects will receive Iloperidone.
  Interventions: Drug: Iloperidone; Drug: Placebo

INTERVENTIONS:
Drug: Iloperidone — Subjects will receive oral iloperidone for 8 weeks. The first 2 weeks of treatment is called titration period and during this time the dose of iloperidone will be increased periodically from 1mg to a maximum of 8mg depending on response and tolerability.
  During the remaining 6 weeks of treatment, called stable dose period, the subjects will receive a stable dose of iloperidone(defined during titration period)
  Other Names: Fanapt; Fanapta; Zomaril
Drug: Placebo — During 8 weeks subjects will receive oral placebo
  Other Names: Sugar pill

SUMMARY:
A Double-Blind Placebo-Controlled Random Order Crossover Pilot Study of Iloperidone for Symptoms of Arousal in PTSD.

DETAILED DESCRIPTION:
During Period A, subjects will receive 8 weeks of iloperidone or placebo (2 weeks titration period followed by 6 weeks on stable dose). Then they will be reassessed for response during Period A; study drug will be discontinued and washed out over the following 2 weeks. They will then begin Period B on the alternate blinded treatment with similar titration and assessment, initially weekly and then every other week for a total of another 8 weeks. The purpose of the study is to determine whether Iloperidone is effective in the treatment of some symptoms in patients with PTSD, particularly difficulty falling or staying asleep, trauma dreams and daytime irritability or outbursts.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis

Exclusion Criteria:

* Pregnancy
* Traumatic Brain Injury greater than mild
* Primary sleep disorder
* Caffeinism
* Active substance use disorder
* Active suicidal risk
* Antipsychotic medication, antibiotics, sedatives, some antihypertensive or antiarrhythmic medication

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Allen, M.D., Principal Investigator — University of Colorado School of Medicine - Depression Center
Locations (1):
- University of Colorado Depression Center; Clinical and Translational Research Center (CTRC), Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Citrome L. Iloperidone for schizophrenia: a review of the efficacy and safety profile for this newly commercialised second-generation antipsychotic. Int J Clin Pract. 2009 Aug;63(8):1237-48. doi: 10.1111/j.1742-1241.2009.02142.x. PMID 19624791
- [Background] David D, De Faria L, Mellman TA. Adjunctive risperidone treatment and sleep symptoms in combat veterans with chronic PTSD. Depress Anxiety. 2006;23(8):489-91. doi: 10.1002/da.20187. PMID 16845653
- [Background] Krystal JH, Rosenheck RA, Cramer JA, Vessicchio JC, Jones KM, Vertrees JE, Horney RA, Huang GD, Stock C; Veterans Affairs Cooperative Study No. 504 Group. Adjunctive risperidone treatment for antidepressant-resistant symptoms of chronic military service-related PTSD: a randomized trial. JAMA. 2011 Aug 3;306(5):493-502. doi: 10.1001/jama.2011.1080. PMID 21813427
- [Background] Kobayashi I, Boarts JM, Delahanty DL. Polysomnographically measured sleep abnormalities in PTSD: a meta-analytic review. Psychophysiology. 2007 Jul;44(4):660-9. doi: 10.1111/j.1469-8986.2007.537.x. Epub 2007 May 22. PMID 17521374
- [Background] Monnelly EP, Ciraulo DA, Knapp C, Keane T. Low-dose risperidone as adjunctive therapy for irritable aggression in posttraumatic stress disorder. J Clin Psychopharmacol. 2003 Apr;23(2):193-6. doi: 10.1097/00004714-200304000-00012. PMID 12640221
- [Background] Raskind MA, Peskind ER, Hoff DJ, Hart KL, Holmes HA, Warren D, Shofer J, O'Connell J, Taylor F, Gross C, Rohde K, McFall ME. A parallel group placebo controlled study of prazosin for trauma nightmares and sleep disturbance in combat veterans with post-traumatic stress disorder. Biol Psychiatry. 2007 Apr 15;61(8):928-34. doi: 10.1016/j.biopsych.2006.06.032. Epub 2006 Oct 25. PMID 17069768
- [Background] Reich DB, Winternitz S, Hennen J, Watts T, Stanculescu C. A preliminary study of risperidone in the treatment of posttraumatic stress disorder related to childhood abuse in women. J Clin Psychiatry. 2004 Dec;65(12):1601-6. doi: 10.4088/jcp.v65n1204. PMID 15641864
- [Background] Taylor FB, Martin P, Thompson C, Williams J, Mellman TA, Gross C, Peskind ER, Raskind MA. Prazosin effects on objective sleep measures and clinical symptoms in civilian trauma posttraumatic stress disorder: a placebo-controlled study. Biol Psychiatry. 2008 Mar 15;63(6):629-32. doi: 10.1016/j.biopsych.2007.07.001. Epub 2007 Sep 14. PMID 17868655
- [Background] Wicklow A, Espie CA. Intrusive thoughts and their relationship to actigraphic measurement of sleep: towards a cognitive model of insomnia. Behav Res Ther. 2000 Jul;38(7):679-93. doi: 10.1016/s0005-7967(99)00136-9. PMID 10875190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single participant was enrolled but did not complete the study.
Groups:
- Iloperidone / Placebo: During 1st treatment period subjects will receive iloperidone. During 2nd treatment period subjects will receive placebo.
  Iloperidone: Subjects will receive oral iloperidone for 8 weeks. The first 2 weeks of treatment is called titration period and during this time the dose of iloperidone will be increased periodically from 1mg to a maximum of 8mg depending on response and tolerability.
  During the remaining 6 weeks of treatment, called stable dose period, the subjects will receive a stable dose of iloperidone(defined during titration period)
  Placebo: During 8 weeks subjects will receive oral placebo
- Placebo / Iloperidone: During 1st treatment period subjects will receive placebo. During 2nd treatment period subjects will receive Iloperidone.
  Iloperidone: Subjects will receive oral iloperidone for 8 weeks. The first 2 weeks of treatment is called titration period and during this time the dose of iloperidone will be increased periodically from 1mg to a maximum of 8mg depending on response and tolerability.
  During the remaining 6 weeks of treatment, called stable dose period, the subjects will receive a stable dose of iloperidone(defined during titration period)
  Placebo: During 8 weeks subjects will receive oral placebo
Period: First Treatment
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Treatment
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Demographics information is not reported for the single study participant to protect confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Administered PTSD Scale (CAPS) Part B and D
Description: The Clinician-Administered PTSD Scale (CAPS) is a structured interview used to diagnose and assess PTSD. Part B of CAPS evaluates symptoms of re-experiencing. Part D evaluates avoidance and numbing.
  CAPS-B scores range from 0 to 40 where higher scores indicate more symptoms. A score 0 means no re-experiencing symptoms.
  CAPS-D scores range form 0 to 56 and higher scores indicate more symptoms. A score 0 means no avoidance or numbing symptoms.
  The primary endpoint was changes in CAPS part B and D after 8 weeks of treatment.
Time Frame: Randomization and at the end of each treatment period. Placebo treatment lasted 8 weeks. Iloperidone treatment lasted 2 weeks.
Population: Study was terminated due to lack of enrollment.
Measure: Number; unit: units on a scale
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Number analyzed (Participants) | 0 | 1
units on a scale
  CAPS part B at randomization 1 |  | 20
  CAPS part B after 8 weeks with placebo |  | 4
  CAPS part B at randomization 2 |  | 4
  CAPS part B after 2 weeks with iloperidone |  | 0
  CAPS part D at randomization 1 |  | 6
  CAPS part D after 8 weeks with placebo |  | 2
  CAPS part D at randomization 2 |  | 7
  CAPS part D after 2 weeks with iloperidone |  | 0

2. Secondary Outcome: Number of Awakenings
Description: Number of awakenings was measured by wrist actigraphy and sleep logs. Actigraphy results were downloaded at each study visit. The mean value during placebo treatment was calculated. There was only 1 value during iloperidone treatment.
Time Frame: Randomization and after 1, 2, 4, 6 and 8 weeks of placebo treatment. Only 1 week of wrist actigraphy was recorded during iloperidone treatment .
Population: Study was terminated due to lack of enrollment. No data for this outcome measure was collected for the single participant.
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Aggression
Description: Aggression was measured by the Modified Overt Aggression Scale (MOAS).This assessment measures four types of aggressive behavior (verbal, aggression against property, autoaggression, and physical aggression) . Total scores on the MOAS range from 0-40, with a higher score indicating more aggressive behavior.
Time Frame: Randomization and 8 weeks of treatment, during both treatment periods
Population: Study was terminated due to lack of enrollment. No data for this outcome measure was collected for the Iloperidone / Placebo arm.
Measure: Number; unit: units on a scale
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Number analyzed (Participants) | 0 | 1
units on a scale
  MOAS at randomization 1 |  | 1
  MOAS after 8 weeks with placebo |  | 0
  MOAS at randomization 2 |  | 0
  MOAS after 2 weeks with iloperidone treatment |  | 0

4. Secondary Outcome: Sleep Latency
Description: Sleep latency was measured by wrist actigraphy and sleep logs. Actigraphy results were downloaded at each study visit. The mean value during placebo treatment was calculated.There was only 1 value during iloperidone treatment
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Wake-time After Sleep Onset (WASO)
Description: WASO was measured by wrist actigraphy and sleep logs. Actigraphy results were downloaded at each study visit. The mean value during placebo treatment was calculated.There was only 1 value during iloperidone treatment.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Suicidal Ideation
Description: The presence of suicidal ideation was monitored over the course of the trial by the first section of the Columbia Suicide Severity Rating Scale (CSSRS). This first section of the scale consists of 5 questions that can be answered yes or no. The number of participants who reported experiencing suicidal ideation is reported.
Time Frame: Total course of the study. CSSRS was administered during each study visit. Suicidal ideation during lifetime and during the month prior to screening were also explored
Population: Study was terminated early due to lack of enrollment.
Measure: Number; unit: participants
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Number analyzed (Participants) | 0 | 1
participants
  Lifetime suicidal ideation |  | 1
  1 month prior to screening |  | 0
  Suicidal ideation during the study |  | 0

7. Secondary Outcome: Intensity of Suicidal Ideation
Description: Intensity of Suicidal Ideation was monitored over the course of the trial by the second section of the Columbia Suicide Severity Rating Scale (CSSRS). This section is only administered if the patient answers yes to the first section. The section consists of 5 questions that refer to the most severe level of ideation endorsed in the first section of the CSSRS. The total score ranges from 2 to 25, with a higher number indicating more intense ideation and greater risk.
  Only lifetime intensity of suicidal ideation was explored as the patient had no suicidal ideation from the month prior to beginning the study to the completion of the study
Time Frame: Baseline
Population: Study was terminated early due to lack of enrollment.
Measure: Number; unit: score on a scale
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Number analyzed (Participants) | 0 | 1
score on a scale |  | 16

8. Secondary Outcome: Suicidal Behavior
Description: The presence and severity os suicidal behavior was monitored over the course of the trial by the third section of the Columbia Suicide Severity Rating Scale (CSSRS). This sections consists of questions about 5 suicidal behaviors and non-suicidal self injurious behavior and it can be answered yes or no. The number of participants who experienced suicidal behavior is reported.
Time Frame: as for outcome 6
Population: Study was terminated due to lack of enrollment.
Measure: Number; unit: participants
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
Number analyzed (Participants) | 0 | 1
participants
  Lifetime suicidal behavior |  | 0
  1 month prior ro screening |  | 0
  During the course of the study |  | 0

ADVERSE EVENTS:
Description: Study was terminated due to lack of enrollment. No participants were enrolled in the "Iloperidone / Placebo" arm
Arm/Group | Iloperidone / Placebo | Placebo / Iloperidone
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No